CLINICAL TRIAL: NCT05462106
Title: A Phase 1b/2, Multicenter, Adaptive, Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Immunogenicity, and Pharmacodynamic Effects of ACI-24.060 in Subjects With Prodromal Alzheimer's Disease and in Adults With Down Syndrome (ABATE)
Brief Title: A Study to Assess the Effects of ACI-24.060 in Alzheimer's Disease and in Down Syndrome (ABATE Study)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AC Immune SA (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ACI-24-AD-DS-2102; 2021-006195-17 (EudraCT Number); 2022-500069-29-00 (Other: European Union Drug Regulatory Authorities Clinical Trial System)
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Amyloid Plaque; Beta-Amyloid; DSAD; Prodromal Alzheimer's Disease; Alzheimer's Disease
Keywords: Dementia; Brain Diseases; Central Nervous System Diseases; Amyloid Plaque; Beta-Amyloid; Down syndrome; Immunogenicity; active immunotherapy; immune response; anti-amyloid therapy; DSAD; Alzheimer's disease
MeSH Terms: conditions — Plaque, Amyloid; Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Placebo for Study Part 1 (Prodromal AD) (Placebo Comparator): Prodromal AD participants receive placebo at predefined time points over 48 weeks
  Interventions: Biological: Placebo
- ACI-24.060 at Dose A in Prodromal AD (Experimental): Prodromal AD participants receive dose A of ACI-24.060 at predefined time points over 48 weeks
  Interventions: Biological: ACI-24.060 at Dose A
- ACI-24.060 at Dose B in Prodromal AD (Experimental): Prodromal AD participants receive dose B of ACI-24.060 at predefined time points over 48 weeks.
  Interventions: Biological: ACI-24.060 at Dose B
- ACI-24.060 at Dose C in Prodromal AD (Experimental): Prodromal AD participants receive dose C of ACI-24.060 at predefined time points over 48 weeks.
  Interventions: Biological: ACI-24.060 at Dose C
- ACI-24.060 at Dose D in Prodromal AD (Optional) (Experimental): Prodromal AD participants receive dose D of ACI-24.060 at predefined time points over 48 weeks. This arm is optional.
  Interventions: Biological: ACI-24.060 at Dose D
- Placebo for Study Part 2 (Down syndrome) (Placebo Comparator): Participants with Down syndrome receive placebo at predefined time points over 74 weeks
  Interventions: Biological: Placebo
- ACI-24.060 at Dose A in Down syndrome (Experimental): Participants with Down syndrome receive dose A of ACI-24.060 at predefined time points over 74 weeks. Dose A will be a dose already tested in Study Part 1.
  Interventions: Biological: ACI-24.060 at Dose A
- ACI-24.060 at Dose B in Down syndrome (Experimental): Participants with Down syndrome may optionally receive a dose B of ACI-24.060 at predefined time points over 74 weeks.
  Interventions: Biological: ACI-24.060 at Dose B
- ACI-24.060 at Dose C in Down syndrome (Experimental): Participants with Down syndrome receive dose C of ACI-24.060 at predefined time points over 74 weeks. Dose C will be a dose already tested in Study Part 1.
  Interventions: Biological: ACI-24.060 at Dose C

INTERVENTIONS:
Biological: Placebo — Administration of Placebo
  Arms: Placebo for Study Part 1 (Prodromal AD)
Biological: ACI-24.060 at Dose A — Administration of Dose A of ACI-24.060
  Arms: ACI-24.060 at Dose A in Prodromal AD
Biological: ACI-24.060 at Dose B — Administration of Dose B of ACI-24.060
  Arms: ACI-24.060 at Dose B in Prodromal AD
Biological: ACI-24.060 at Dose C — Administration of Dose C of ACI-24.060
  Arms: ACI-24.060 at Dose C in Prodromal AD
Biological: ACI-24.060 at Dose D — Administration of Dose D of ACI-24.060
  Arms: ACI-24.060 at Dose D in Prodromal AD (Optional)
Biological: Placebo — Administration of Placebo
  Arms: Placebo for Study Part 2 (Down syndrome)
Biological: ACI-24.060 at Dose A — Administration of Dose A of ACI-24.060. Dose A will be a dose already tested in Study Part 1
  Arms: ACI-24.060 at Dose A in Down syndrome
Biological: ACI-24.060 at Dose B — Administration of Dose B of ACI-24.060
  Arms: ACI-24.060 at Dose B in Down syndrome
Biological: ACI-24.060 at Dose C — Administration of Dose C of ACI-24.060
  Arms: ACI-24.060 at Dose C in Down syndrome

SUMMARY:
The purpose of this study is to assess the safety, tolerability, immunogenicity and pharmacodynamic effects of ACI-24.060 in subjects with prodromal Alzheimer's disease and in non-demented adults with Down syndrome.

DETAILED DESCRIPTION:
This phase 1b/2 study will be in 2 parts. Study Part 1 will involve subjects with prodromal Alzheimer's disease. Study Part 2 will involve subjects with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

Study Part 1

1. Age ≥50 and ≤85 years at screening.
2. Diagnosis of prodromal AD: MCI due to AD according to National Institute on Aging Alzheimer's Association (NIA-AA) criteria.
3. PET scan at screening consistent with the presence of amyloid pathology.
4. Clinical Dementia Rating (CDR)-Global Score of 0.5.
5. Subjects either not taking any marketed treatment for AD or receiving a stable dose of an acetylcholinesterase inhibitor (ACHEI) and/or memantine for at least 2 months prior to baseline.

Study Part 2

1. Age ≥35 and ≤50 years at screening (subjects with DS with age ≥35 and ≤39 years may be considered on the condition that there is prior evidence of amyloid results compatible with AD pathology at PET-scan and/or in biofluids).
2. Male or female subjects with DS with a cytogenetic diagnosis being either trisomy 21 or complete unbalanced translocation of the chromosome 21.
3. PET scan at screening consistent with the presence of amyloid pathology.
4. Mild to moderate intellectual disability as per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) classification.
5. Subjects must have a study partner who has direct and regular contact, at least 10 hours per week, with the subject and who is able to provide reliable answers to questions related to the subject, according to the study investigator.

Exclusion Criteria:

1. Any unstable and/or clinically significant medical condition likely to hamper the evaluation of safety and/or efficacy of the study treatment (eg, moderate and/or severe untreated obstructive sleep apnea, clinically significant reduction in serum B12 or folate levels, clinically significant abnormalities of thyroid function, stroke, or other cerebrovascular conditions), as per investigator's judgement.
2. DSM-5 criteria for drug or alcohol abuse or dependence currently met within the past 5 years.
3. History or presence of uncontrolled seizures. If history of seizures, they must be well controlled with no occurrence of seizures in the 2 years before study screening. The use of antiepileptic medications is permitted.
4. Concomitant or past history psychiatric or neurologic disorder other than those considered to be related to AD (eg, head injury with loss of consciousness, symptomatic stroke, Parkinson's disease, severe carotid occlusive disease, transient ischemic attacks [TIAs], hemorrhagic and/or non-hemorrhagic stroke).
5. History of meningitis or meningoencephalitis.
6. History of moderate or severe traumatic brain injury.
7. History of or presence of inflammatory neurological disorders.
8. History or presence of immunological or autoimmune disorders.
9. History of severe allergic reaction (eg, anaphylaxis) including, but not limited to severe allergic reaction to previous vaccines, foods, and/or medications.
10. Significant risk of suicide, defined using the C-SSRS as the subject answering "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior within the past 12 months.
11. MRI scan at screening showing a single area of cerebral vasogenic edema, superficial siderosis, or evidence of a previous macro-hemorrhage or showing more than 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"). Evidence of space occupying lesions other than benign meningioma of less than 1 cm diameter, more than 2 lacunar infarcts, or 1 single infarct larger than 1 cm in diameter. Screening MRI scan showing structural evidence of alternative pathology not consistent with AD and is considered to be at the origin of subject's symptoms.
12. Deviations from normal values for hematologic parameters, liver function tests, and other biochemical measures, judged to be clinically significant by the investigator.
13. Subjects with a positive Human Immunodeficiency Virus (HIV-1 and 2) test at screening.
14. Subjects with clinical or laboratory evidence of active hepatitis B or C at screening (eg, HBV or HCV antigens).
15. Subjects with positive syphilis serology consistent with active syphilis at screening.
16. Subjects with presence of antibody titers related to immunological or autoimmune disorders at screening.
17. MRI examination cannot be done for any reason, including but not limited to metal implants contraindicated for MRI and/or severe claustrophobia.
18. Any contraindication for PET scan imaging.
19. Any contraindication to lumbar puncture in subjects undergoing this procedure (note: lumbar puncture is optional in subjects with DS).
20. Previous treatment with ACI-24 or any other active immunotherapy against AD at any time in the past unless there is firm evidence that the subject received placebo only and the placebo formulation is not expected to induce any specific immune response.
21. Previous treatment with any investigational and/or marketed passive immunotherapy against AD within 6 months before screening or 5 half-lives, whichever is longer, unless there is firm evidence that the subject received placebo only.
22. Ongoing treatment with any approved anti-amyloid passive immunotherapy for Alzheimer's disease.
23. Use of acetylcholinesterase inhibitor or glutamatergic drugs (eg, memantine, topiramate, lamotrigine) if not on stable dose for at least 2 months before screening.
24. Any vaccine, either live or not, including but not limited to influenza or COVID-19 vaccine, received within 4 weeks before randomization.
25. Subjects with treated hypothyroidism not on a stable dose of replacement medication for at least 2 months before screening and having clinically significant abnormal serum T4 and/or thyroid stimulating hormone at screening.
26. Subjects undergoing lumbar puncture and being treated with any anticoagulants or antiplatelet drugs, except aspirin at doses of 100 mg daily or lower.
27. Use of antidepressants (other than selective serotonin reuptake inhibitors/serotonin-norepinephrine reuptake inhibitors at stable dose); typical antipsychotics; γ-aminobutyric acid agonists (eg, gabapentin); or stimulants (eg, methylphenidate, modafinil). Stable doses of atypical antipsychotics or benzodiazepines are only allowed if this is not considered to influence the safety and the efficacy of the study treatment according to the site investigator and the sponsor medical monitor.
28. Chronic use of opioid analgesics. A limited treatment duration for acute conditions until 24 hours before cognitive assessment is allowed.
29. Current use of immunosuppressant or immunomodulating drugs or their use within the 6 months before study screening. Current use of oral steroids or their use within the 3 months before study screening.

    Additional Exclusion Criteria in Study Part 2

    The following are exclusion criteria at the time of randomization but will not be considered as exclusionary after treatment assignment:
30. Clinical diagnosis of AD dementia in DS as per International Classification of Diseases 10 (ICD-10).
31. DSQIID >20.
32. Intelligence quotient score <40 (KBIT-2).

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) assessed by intensity (mild, moderate or severe) and causal relationship (unrelated, unlikely, possibly or probably related) | From Screening to Week 74 (Study Part 1)
Number of participants with Adverse Events (AEs) assessed by intensity (mild, moderate or severe) and causal relationship (unrelated, unlikely, possibly or probably related) | From Screening to Week 100 (Study Part 2)
Number of participants with abnormal MRI results | From Baseline to Week 74 (Study Part 1)
Number of participants with abnormal MRI results | From Baseline to Week 100 (Study Part 2)
Number of participants with abnormal physical and neurological examination results | From Baseline to Week 74 (Study Part 1)
Number of participants with abnormal physical and neurological examination results | From Baseline to Week 100 (Study Part 2)
Number of participants reporting suicidal ideation or behavior using Columbia-Suicide Severity Rating Scale (C-SSRS) | From Baseline to Week 74 (Study Part 1)
Number of participants reporting suicidal ideation or behavior using Columbia-Suicide Severity Rating Scale (C-SSRS) | From Baseline to Week 100 (Study Part 2)
Change from baseline in Anti-Abeta antibody titers in blood | From Baseline to Week 100 (Study Part 2)

SECONDARY OUTCOMES:
Change from baseline in Anti-Abeta antibody titers | From Baseline to Week 74 (Study Part 1)
Change from baseline on brain amyloid levels | From Baseline to W100 (Study Part 2)
  Brain amyloid load measured via PET imaging. An increase indicates a worsening.

OTHER OUTCOMES:
Change from baseline on brain amyloid levels | From Baseline to W48 (Study Part 1)
  Brain amyloid load measured via PET imaging. An increase indicates a worsening.
Change from baseline on tau levels | From Baseline to W48 (Study Part 1) and to W100 (Study Part 2)
  Brain tau load measured via PET imaging. An increase indicates a worsening.
Change from baseline in cognitive tests - Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | From Baseline to Week 74 (Study Part 1)
  The total scale index score ranges from 40 to 160. A higher score indicates a better outcome.
Change from baseline in cognitive tests - Alzheimer's Disease Assessment Scale-Cognitive Subscale 13 item (ADAS-Cog 13) | From Baseline to Week 74 (Study Part 1)
  The score ranges from 0 to 85. A higher score indicates a worse outcome.
Change from baseline in clinical function tests - Clinical Dementia Rating Scale (CDR) | From Baseline to Week 74 (Study Part 1)
  The score ranges from 0 to 18. A higher score indicates a worse outcome.
Change from baseline in cognitive tests - Modified Cued Recall Test (mCRT) | From Baseline to Week 100 (Study Part 2)
  The modified CRT assesses verbal learning and episodic memory. The score ranges from X to Y. A higher score indicates a better outcome.
Change from baseline in cognitive tests - Cambridge Cognitive Examination for Individuals with Down Syndrome (CAMCOG-DS2) | From Baseline to Week 100 (Study Part 2)
  CAMCOG-DS measures cognitive decline. The total score ranges from 0 to 107. A higher score indicates a better outcome.
Change from baseline in cognitive tests - Cambridge Neuropsychological Test Automated Battery-Paired Associates Learning (CANTAB-PAL) | From Baseline to Week 100 (Study Part 2)
  The CANTAB-PAL assesses visual memory and new learning. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rafii, MD, Principal Investigator — University of Southern California, Alzheimer's Therapeutic Research Institute, 9860 Mesa Rim Rd, San Diego, CA 92121, USA
Locations (19):
- United States (7):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Indiana University / IU Health, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Fairway, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Washington University, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Health San Antonio, San Antonio, Texas
- Spain (7):
  - Fundació ACE, Institut Català de Neurociències Aplicades, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen De Las Nieves, Granada
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (5):
  - Cambridge and Peterborough NHS Foundation Trust - Windsor Research Units, Cambridge
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Re:Cognition Health Limited, London
  - South London and Maudsley NHS Foundation Trust of The Maudsley Hospital, London
  - Oxford Health NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Undecided